CLINICAL TRIAL: NCT04014829
Title: Evaluation of Central Sensitization, Fear-Avoidance, and Pain-Pressure Threshold With Chronic Pain in Post-Hysterectomy Patients: A Collaborative Cohort Study (EPOCH - Enhancing Post-operative Outcomes in Chronic Pain After Hysterectomy)
Brief Title: Evaluation of Central Sensitization, Fear-Avoidance, and Pain-Pressure Threshold With Chronic Pain After Hysterectomy
Acronym: EPOCH
Status: Recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: EPOCH
Record Dates: First submitted 2019-07-05; First posted 2019-07-10 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hysterectomy; Chronic Pain; Central Sensitisation; Anxiety Depression
Keywords: Hysterectomy; Chronic Pain; Fear-Avoidance; Central Sensitization; Pain-Pressure Threshold; Mechanical Temporal Summation; Heart rate variability
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group for CPHP: Preoperative assessment with questionnaires, Mechanical Temporal Summation, Pain-Pressure Threshold, and heart rate variability. All patients will undergo elective abdominal or laparoscopic hysterectomy. Patients will be assigned to this group if no significant pain is noted during the follow up evaluations at 4 and 6 months.
  Interventions: Diagnostic Test: Pain-Pressure Threshold; Diagnostic Test: Mechanical Temporal Summation; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Pain Catastrophizing Scale; Diagnostic Test: Central Sensitization Inventory; Diagnostic Test: Fear-Avoidance Component Score; Diagnostic Test: EQ-5D; Diagnostic Test: heart rate variability; Diagnostic Test: Anxiety, anticipated pain, anticipated analgesia; Diagnostic Test: State-trait anxiety inventory; Diagnostic Test: Beck's Depression Inventory
- Chronic Post-Hysterectomy Pain (CPHP): Preoperative assessment with questionnaires, Mechanical Temporal Summation, Pain-Pressure Threshold, and heart rate variability. All patients will undergo elective abdominal or laparoscopic hysterectomy. Patients will be assigned to this group if significant pain is noted during the follow up evaluations at 4 and 6 months.
  Interventions: Diagnostic Test: Pain-Pressure Threshold; Diagnostic Test: Mechanical Temporal Summation; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Pain Catastrophizing Scale; Diagnostic Test: Central Sensitization Inventory; Diagnostic Test: Fear-Avoidance Component Score; Diagnostic Test: EQ-5D; Diagnostic Test: heart rate variability; Diagnostic Test: Anxiety, anticipated pain, anticipated analgesia; Diagnostic Test: State-trait anxiety inventory; Diagnostic Test: Beck's Depression Inventory
- Control group for significant postoperative pain: Preoperative assessment with questionnaires, Mechanical Temporal Summation, Pain-Pressure Threshold, and heart rate variability. All patients will undergo elective abdominal or laparoscopic hysterectomy. Patients will be assigned to this group if no significant pain is noted during the follow up evaluations at 24 and 48 hours.
  Interventions: Diagnostic Test: Pain-Pressure Threshold; Diagnostic Test: Mechanical Temporal Summation; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Pain Catastrophizing Scale; Diagnostic Test: Central Sensitization Inventory; Diagnostic Test: Fear-Avoidance Component Score; Diagnostic Test: EQ-5D; Diagnostic Test: heart rate variability; Diagnostic Test: Anxiety, anticipated pain, anticipated analgesia; Diagnostic Test: State-trait anxiety inventory; Diagnostic Test: Beck's Depression Inventory
- Significant postoperative pain: Preoperative assessment with questionnaires, Mechanical Temporal Summation, Pain-Pressure Threshold, and heart rate variability. All patients will undergo elective abdominal or laparoscopic hysterectomy. Patients will be assigned to this group if significant pain is noted during the follow up evaluations at 24 and 48 hours.
  Interventions: Diagnostic Test: Pain-Pressure Threshold; Diagnostic Test: Mechanical Temporal Summation; Diagnostic Test: Hospital Anxiety and Depression Scale; Diagnostic Test: Pain Catastrophizing Scale; Diagnostic Test: Central Sensitization Inventory; Diagnostic Test: Fear-Avoidance Component Score; Diagnostic Test: EQ-5D; Diagnostic Test: heart rate variability; Diagnostic Test: Anxiety, anticipated pain, anticipated analgesia; Diagnostic Test: State-trait anxiety inventory; Diagnostic Test: Beck's Depression Inventory

INTERVENTIONS:
Diagnostic Test: Pain-Pressure Threshold — Performed on bilateral trapezius muscles. Pressure will be applied at 90 degrees downward with an algometer, with the speed of pressure increase approximately 1kgf/s. Upon the sensation of pain, the patient will vocalize or raise her hand to terminate the test, and the highest reading will be recorded (up to maximum 6kgf). If two values are recorded within 0.2kgf of each other, the mean value will be recorded. If two values are greater than 0.2kgf of each other, a third test will be performed and the mean obtained.
  Other Names: PPT
Diagnostic Test: Mechanical Temporal Summation — Pinprick hyperalgesia will be evoked using a Von Frey filament, applied to the volar aspect of the dominant forearm. Participants will report using the numerical rating scale the intensity of pain from the first stimulus. Subsequently, ten repetitive stimuli one second apart will be applied with the same filament within an area of 1cm diameter of the same forearm. Subjects will report the rate the pain intensity of the tenth stimulus. The magnitude of MTS is calculated as the difference between the last to the first pain scores. The investigators will classify the participants according to "evoked MTS" if the last stimulus is rated higher than the first, or "no MTS" if the last stimulus is rated equal or lower than the first. The research team administering the test will follow a set script.
  Other Names: MTS
Diagnostic Test: Hospital Anxiety and Depression Scale — Standardized questionnaire to determine the level of anxiety and depression.
  Other Names: HADS
Diagnostic Test: Pain Catastrophizing Scale — Standardized questionnaire to determine the level of pain catastrophizing.
  Other Names: PCS
Diagnostic Test: Central Sensitization Inventory — Standardized questionnaire to determine the level of central sensitization.
  Other Names: CSI
Diagnostic Test: Fear-Avoidance Component Score — Standardized questionnaire to determine the level of fear and avoidance.
  Other Names: FACS
Diagnostic Test: EQ-5D — Standardized questionnaire to assess generic health-related quality of life.
Diagnostic Test: heart rate variability — Heart rate variability will be determined from the R-to-R intervals obtained from a 5-minute ECG recording.
  Other Names: HRV
Diagnostic Test: Anxiety, anticipated pain, anticipated analgesia — Preoperative anxiety (0 to 100), anticipated pain (0 to 100), and anticipated analgesia requirement (0 to 5).
Diagnostic Test: State-trait anxiety inventory — Standardized questionnaire to assess anxiety.
  Other Names: STAI
Diagnostic Test: Beck's Depression Inventory — Standardized questionnaire to assess depressive symptoms.
  Other Names: BDI

SUMMARY:
Phase 1 (started in July 2019):

Central Sensitization Inventory (CSI), Fear-Avoidance Components Scale (FACS), pain-pressure threshold are factors associated with chronic post-hysterectomy pain (CPHP), but a complete understanding on the development of CPHP is lacking. The study aims to identify clinically-relevant factors for CPHP that can be reliably assessed preoperatively.

===

Phase 2 (anticipated start May 2022):

In addition to above factors, the association between heart rate variability (HRV) parameters, anxiety level, anticipated pain, and anticipated analgesia requirement with significant postoperative pain and CPHP will be investigated.

DETAILED DESCRIPTION:
Phase 1 (started in July 2019):

Chronic post-surgical pain is persistent pain after a surgical procedure that lasts for at least 3 months with other causes of pain excluded. It is a major socioeconomic and healthcare burden, and has impact on quality of life, physical function, emotional wellbeing and healthcare costs. In Singapore, hysterectomy for benign indications incurs 32% risk of developing chronic post-hysterectomy pain (CPHP). CPHP can occur around the surgical site, lower abdominal or pelvic region. Based on the pathophysiology underlying chronic pain, the investigators hypothesize that central sensitization, pain fear-avoidance and low pain-pressure threshold are plausible risk factors for CPHP. However, none of these three risk categories has been evaluated in patients with CPHP.

The investigators hypothesize that preoperatively abnormal central sensitization, pain fear-avoidance and decreased pain-pressure threshold are associated with increased risk of developing CPHP. The investigators will evaluate these risk factors preoperatively, and follow-up study participants at 4- and 6-months after hysterectomy, to assess the associations between these risk factors and CPHP.

The investigators will perform a prospective study of 236 patients undergoing abdominal/laparoscopic hysterectomy for benign indications, recruited at KK Hospital, Singapore. Central Sensitization Inventory (CSI), Fear-Avoidance Components Scale (FACS), pain-pressure threshold and other known factors associated with CPHP will be assessed and recorded. Participants will be followed up at 4- and 6-months postoperatively to assess CPHP. Logistical regression analysis will be used to evaluate the associations between these factors and CPHP.

Knowledge of risk factors for CPHP will guide future studies to identify high-risk patients for implementation of individualized targeted therapies to optimize surgical outcomes of this patient group, and to confirm the hypothetical pathophysiological processes of chronic post-surgical pain similarly applicable to CPHP.

===

Phase 2 (anticipated start May 2022):

Recent evidence suggests that changes in heart rate variability (HRV) parameters, anxiety level, anticipated pain, and anticipated analgesia requirement may be associated with significant postoperative pain (numerical pain score >3 out of 10). The associations between HRV, anxiety level, anticipated pain, and anticipated analgesia requirement with significant pain or CPHP after hysterectomy have yet been investigated.

The investigators hypothesize that preoperative changes in HRV parameters, increased anxiety level, higher anticipated pain, and higher anticipated analgesia requirement are associated with increased risk of developing significant postoperative pain or CPHP. HRV, anxiety level, anticipated pain, and anticipated analgesia requirement will be assessed preoperatively, and follow-up study participants at 24 hours, 48 hours, 4- and 6-months after hysterectomy to assess their associations with significant postoperative pain and CPHP.

The investigators will perform a prospective study of 200 patients undergoing abdominal/laparoscopic hysterectomy for benign indications, recruited at KK Hospital, Singapore. HRV, anxiety level, anticipated pain, and anticipated analgesia requirement will be assessed and recorded. Participants will be followed up at 24 hours, 48 hours, 4- and 6-months postoperatively to assess significant pain and CPHP. Logistical regression analysis will be used to evaluate the associations between these factors and significant pain or CPHP.

Knowledge of risk factors for significant pain and CPHP will guide future studies to identify high-risk patients for implementation of individualized targeted therapies to optimize surgical outcomes of this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 80 years old
* American Society of Anesthesiologists Physical Scale (ASA) I to III
* Benign gynaecological indications for hysterectomy
* Elective abdominal or laparoscopic hysterectomy

Exclusion Criteria:

* Vaginal hysterectomy
* Uterine prolapse, endometriosis, malignant disease, or pelvic pain as main indication for surgery
* History of drug dependence or recreational drug use
* History of chronic pain syndrome
* Current chronic daily treatment with corticosteroids, excluding inhaled steroids
* Allergy to study drugs
* Major heart surgery
* Heart transplant
* Pacemaker inserted
* Baseline non-sinus cardiac rhythm

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysterectomy is a surgical procedure that is performed only on women
Study Population: Women scheduled for elective abdominal or laparoscopic hysterectomy at KK Women's and Children's Hospital, Singapore.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Chronic Post-Hysterectomy Pain at 4 months | 4 months after hysterectomy
  The primary outcome measure is the development of chronic post-hysterectomy pain, which is defined as pain that lasts for at least 3 months around the surgical site, lower abdominal, or pelvic region. This will be determined by phone or online assessment at 4 months after surgery, based on the protocol used by Brandsborg et al and the investigators' previous study.
Significant postoperative pain at 24 hours | 24 hours after hysterectomy
  Numerical pain score (0: no pain; 100: worst pain imaginable) will be assessed at 24 hours after hysterectomy with patient moving from supine to sitting position.

SECONDARY OUTCOMES:
Central Sensitization Inventory (CSI) | 2 months (upon recruitment until before surgery)
  Assessment via the validated Central Sensitization Inventory (CSI) questionnaire prior to hysterectomy. Central sensitization is defined as an increased responsiveness of nociceptive neurons in the central nervous system to normal or sub-threshold afferent stimuli. The CSI a 25-item questionnaire, with each item rated 0 to 4. A higher value indicates greater central sensitization, and a threshold score of 40 was shown to be associated with increased risk of chronic pain.
Fear Avoidance Components Scale (FACS) | 2 months (upon recruitment until before surgery)
  Assessment via the validated Fear Avoidance Components Scale (FACS) questionnaire prior to hysterectomy. Fear-avoidance is defined as the negative emotional perception of pain as terrorizing, which can generate catastrophic thoughts and vigilance. Pain fear-avoidance behavior can be assessed with the FACS, a 20-item questionnaire, with each item rated 0 to 5.
Hospital Anxiety and Depression Scale (HADS) | 2 months (upon recruitment until before surgery)
  Assessment via the validated Hospital Anxiety and Depression Scale (HADS) questionnaire prior to hysterectomy. Anxiety and depression are known risk factors associated with CPHP. HADS is a combination test for both anxiety and depression, is a 14-item questionnaire, with each item rated 0 to 3. HADS > 8 has been associated specifically with increased CPHP.
Pain Catastrophizing Scale (PCS) | 2 months (upon recruitment until before surgery)
  Assessment via the validated Pain Catastrophizing Scale (PCS) questionnaire prior to hysterectomy. Pain catastrophizing refers to the negative thought processes patients have when they are exposed to pain or painful experiences. The PCS is a 13-item scale, with each item rated on a 5-point scale: 0 (Not at all) to 4 (all the time). It is broken into three subscales being magnification (0-12), rumination (0-16), and helplessness (0-24). A higher value in each subscale indicates a higher tendency to that subscale (worse outcome).
Quality of life via EQ-5D | 2 months (upon recruitment until before surgery)
  Assessment via the validated EQ-5D questionnaire prior to hysterectomy. Lower preoperative quality of life has been associated with CPHP. EQ-5D is a validated questionnaire to assess generic health-related quality of life, consisting of two components: health state description and evaluation.
  The description component measures health status via five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with each dimension rated according to severity using a three-level scale.
  The evaluation component assesses overall health status using the visual analogue scale (EQ-VAS).
Mechanical Temporal Summation (MTS) | 2 months (upon recruitment until before surgery)
  Assessment via Mechanical Temporal Summation before hysterectomy. A 180 gram von Frey filament is applied on the subject's forearm. Patient will then be asked to rate the pinprick pain score on a verbal rating scale, 0-100. Following this, 10 consecutive touches at random locations are applied with a 1 second interstimulus interval and within a 1 cm diameter circle. The patient will then be asked to rate the 10th pain score (0-100). The Mechanical Temporal Summation Score is obtained by the difference between the 11th pain score and the 1st pain score. If the score is greater than zero, the patient is implied to have presence of Mechanical Temporal Summation.
Pain-Pressure Threshold (PPT) | 2 months (upon recruitment until before surgery)
  Assessment of Pain-pressure threshold (PPT) prior to hysterectomy. PPT is measured via an algometer in both groups. Pressure is applied 90 degree straight down force on the subject's right/left centre of the trapezius muscle using an algometer, with a speed of pressure ~ 1kgf/s. The above procedure is then repeated 3 times at each site (left/right) which is indicated on the pressure mark with each time having the reading recorded. When patient shows no response ≥ 6kgf, the threshold is recorded as 6kgf. The patient upon feeling pain will say stop or raise the hand to terminate the test. The mean value is obtained by averaging the readings and will then be recorded as the threshold estimate.
Chronic Post-Hysterectomy Pain at 6 months | 6 months after hysterectomy
  The primary outcome measure is the development of chronic post-hysterectomy pain, which is defined as pain that lasts for at least 3 months around the surgical site, lower abdominal, or pelvic region. This will be determined by phone or online assessment at 6 months after surgery, based on the protocol used by Brandsborg et al and the investigators' previous study.
heart rate variability | Preoperative and 24 hours after hysterectomy
  Heart rate variability will be determined from the R-to-R intervals obtained from a 5 minute ECG recording with the patient supine.
Preoperative anxiety | Preoperative
  Patients will be asked to rate, using a 0-100 mm visual analog scale (VAS), their surgical anxiety level ("On a scale of 0-100, with 0 being not anxious at all through 100 being extremely anxious, how anxious are you about your upcoming surgery?")
State-Trait Anxiety Inventory | 2 months (upon recruitment until before surgery)
  Assessment via State-Trait Anxiety Inventory questionnaire prior to hysterectomy, a standardized assessment of anxiety. This is a validated 40-item questionnaire, each item scored using a categorical scale from 1-4, with total score from 40 to 160.
Beck's Depression Inventory | 2 months (upon recruitment until before surgery)
  Assessment via Beck's Depression Inventory questionnaire prior to hysterectomy, a standardized assessment of depressive symptoms.This is a validated 21-item questionnaire, each item scored using a categorical scale from 0-3, with total score from 0 to 63.
Anticipated pain | Preoperative
  Patients will be asked to rate, using a 0-100 mm visual analog scale (VAS), their anticipated pain ("On a scale of 0-100, with 0 being no pain at all and 100 being pain as bad as you can imagine, how much pain do you anticipate experiencing after your upcoming surgery?")
Anticipated analgesia requirement | Preoperative
  Patients will be asked to rate, using a categorical scale, their anticipated pain medication need ("On a scale of 0-5, with 0 being none at all, 1 being much less than average, 2 being less than average, 3 being average, 4 being more than average, and 5 being much more than average, how much pain medication do you anticipate needing after your upcoming surgery?")

CONTACTS AND LOCATIONS:
Overall Officials: Farida Ithnin, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapman CR, Vierck CJ. The Transition of Acute Postoperative Pain to Chronic Pain: An Integrative Overview of Research on Mechanisms. J Pain. 2017 Apr;18(4):359.e1-359.e38. doi: 10.1016/j.jpain.2016.11.004. Epub 2016 Nov 28. PMID 27908839
- [Background] Han C, Ge Z, Jiang W, Zhao H, Ma T. Incidence and risk factors of chronic pain following hysterectomy among Southern Jiangsu Chinese Women. BMC Anesthesiol. 2017 Aug 11;17(1):103. doi: 10.1186/s12871-017-0394-3. PMID 28800726
- [Background] Pinto PR, McIntyre T, Nogueira-Silva C, Almeida A, Araujo-Soares V. Risk factors for persistent postsurgical pain in women undergoing hysterectomy due to benign causes: a prospective predictive study. J Pain. 2012 Nov;13(11):1045-57. doi: 10.1016/j.jpain.2012.07.014. Epub 2012 Oct 12. PMID 23063345
- [Background] Sng BL, Ching YY, Han NR, Ithnin FB, Sultana R, Assam PN, Sia ATH. Incidence and association factors for the development of chronic post-hysterectomy pain at 4- and 6-month follow-up: a prospective cohort study. J Pain Res. 2018 Mar 27;11:629-636. doi: 10.2147/JPR.S149102. eCollection 2018. PMID 29628772
- [Background] Fingleton C, Smart K, Moloney N, Fullen BM, Doody C. Pain sensitization in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Jul;23(7):1043-56. doi: 10.1016/j.joca.2015.02.163. Epub 2015 Mar 5. PMID 25749012
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Neblett R, Mayer TG, Hartzell MM, Williams MJ, Gatchel RJ. The Fear-avoidance Components Scale (FACS): Development and Psychometric Evaluation of a New Measure of Pain-related Fear Avoidance. Pain Pract. 2016 Apr;16(4):435-50. doi: 10.1111/papr.12333. Epub 2015 Jul 31. PMID 26228238
- [Background] Brandsborg B, Dueholm M, Kehlet H, Jensen TS, Nikolajsen L. Mechanosensitivity before and after hysterectomy: a prospective study on the prediction of acute and chronic postoperative pain. Br J Anaesth. 2011 Dec;107(6):940-7. doi: 10.1093/bja/aer264. Epub 2011 Sep 2. PMID 21890662

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT04014829/Prot_SAP_000.pdf